CLINICAL TRIAL: NCT02145377
Title: A Phase 2 Randomized, Double-Blinded Study to Compare in Malian Adults the Immunogenicity, Clinical Acceptability and Excretion Pattern Following the Ingestion of a Single Dose of PXVX0200 (CVD 103-HgR) Live Oral Cholera Vaccine Containing Either 108 Colony Forming Units [Cfu] or 109 Cfu Using Shanchol™ Killed Whole Cell Oral Cholera Vaccine as an Immunological Comparator
Brief Title: PXVX0200 (CVD103-HgR) vs Shanchol in Mali
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Emergent BioSolutions (Industry); Shantha Biotechnics Limited (Industry)
Responsible Party: Principal Investigator, Milagritos Tapia, Assistant Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HP-00059690
Record Dates: First submitted 2014-05-20; First posted 2014-05-22 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Cholera
Keywords: Cholera; Vaccine; Mali
MeSH Terms: conditions — Cholera | interventions — shanchol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- PXVX0200 10E8 then placebo (Experimental): PXVX0200 10E8 on day 0; Placebo on day 14
  Interventions: Biological: PXVX0200 10E8; Biological: Placebo
- Placebo, then PXVX0200 10E8 (Experimental): Placebo on day 0; PXVX0200 10E8 on day 14
  Interventions: Biological: PXVX0200 10E8; Biological: Placebo
- PXVX0200 10E9 then Placebo (Experimental): PXVX0200 10E9 on day 0; Placebo on day 14
  Interventions: Biological: PXVX0200 10E9; Biological: Placebo
- Placebo then PXVX0200 10E9 (Experimental): Placebo on day 0; PXVX0200 10E9 on day 14
  Interventions: Biological: PXVX0200 10E9; Biological: Placebo
- Shanchol (Active Comparator): Two doses of Shanchol, on day 0 and day 14
  Interventions: Biological: Shanchol

INTERVENTIONS:
Biological: PXVX0200 10E8 — Oral dose of PXVX0200 10E8
  Arms: PXVX0200 10E8 then placebo; Placebo, then PXVX0200 10E8
Biological: PXVX0200 10E9 — Oral dose of PXVX0200 10E9
  Arms: PXVX0200 10E9 then Placebo; Placebo then PXVX0200 10E9
Biological: Placebo — Oral dose of sodium bicarbonate buffer
  Arms: PXVX0200 10E8 then placebo; PXVX0200 10E9 then Placebo; Placebo then PXVX0200 10E9; Placebo, then PXVX0200 10E8
Biological: Shanchol — Licensed comparator
  Arms: Shanchol

SUMMARY:
To compare the ability of a single dose of PXVX0200 at two different dose levels, to placebo to elicit a significant antibody response 14 days after vaccination, compared to baseline.

To compare the ability of a single dose of PXVX0200 to a comparator vaccine Shanchol, a two dose administration, to elicit antibody response by 14 days after vaccination.

DETAILED DESCRIPTION:
Currently there are two licensed inactivated vibrio oral vaccines (Dukoral® [Crucell; Leiden, The Netherlands] and Shanchol™ [Shantha Biotechnics; Hyderabad, India]) that are pre-qualified by the World Health Organization (WHO) for procurement by United Nations (UN) agencies. Each of these vaccines requires a two-dose regimen which is difficult to implement in the face of explosive outbreaks of cholera in unsettled situations in developing countries. For this reason there is great interest in identifying a cholera vaccine that can provide rapid onset of protection following the ingestion of just a single oral dose.

This Phase 2 randomized, observer-blinded and subject-blinded clinical trial to be conducted in Bamako, Mali will assess the immunogenicity of the 10^8 cfu versus the 10^9 cfu formulation of PaxVax-manufactured CVD 103-HgR.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand the study and give consent (either written or through a process that involves audio tapes explaining all aspects of the study and the consent form in local languages [Bambara and French] followed by making a mark and signature by a literate witness)
* Healthy men or women, age 18 to 45 years (inclusive) without significant medical history
* Women of child-bearing potential must have negative urine pregnancy test at baseline, prior to vaccination. They must also be willing to use adequate birth control for the duration of the 28-day study and have additional pregnancy tests if indicated. Effective methods of birth control for this study include abstinence, intrauterine device (IUD), oral or depot contraceptive, or barrier plus spermicide
* Willingness to remain in the study area until at least 42 days after receipt of the first vaccine dose

Exclusion Criteria:

* Health care workers who have direct contact with patients who are immune deficient, HIV-positive, or have an unstable medical condition
* Clinically significant history of immunodeficiency, cardiovascular disease, respiratory disease, endocrine disorder, liver disease, renal disease, gastrointestinal disease, neurologic illness, psychiatric disorder requiring hospitalization, current drug or alcohol abuse
* History of an abnormal stool pattern or regular use of laxatives
* Previously received a licensed or investigational cholera vaccine
* History of cholera illness

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2014-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
To elicit a significant rise in serum Inaba vibriocidal antibody after a single vaccination | 14 days
  A comparison of the ability of a single ≥2 x10E9 cfu oral dose versus a single ≥2 x10E8 cfu oral dose of PXVX0200 (CVD 103-HgR) versus placebo to elicit a significant (> 4-fold) rise in serum Inaba vibriocidal antibody 14 days after vaccination, compared to baseline

SECONDARY OUTCOMES:
To measure antibody response for a 10E8 dose and 10E9 dose of PXVX0200 oral vaccine | 14 days
  To compare the ability of a single ≥2 x108 cfu dose of PXVX0200 (CVD 103-HgR) or ≥2 x109 oral dose of PXVX0200 (CVD 103-HgR) versus Shanchol™ to elicit serum Inaba vibriocidal antibody mean fold rise (compared to baseline titer) and GMT
To plot the kinetics of the serum Inaba Vibriocidal antibody response | Baseline and post-vaccination time point.
  To plot the kinetics of the serum Inaba vibriocidal antibody response after ingestion of a single oral dose of PXVX0200 (CVD 103-HgR) containing ≥2 x10E8 cfu or ≥2 x10E9 cfu versus Shanchol™. (With GMT on the Y axis and time points on the X axis, the GMTs at baseline and at each post-vaccination time point will be connected as a line graph).
Assess fecal shedding of PXVX0200 | Day 1-3, day 7 and day 14
  Shedding of CVD 103-HgR in stool as determined by stool culture (whole specimen or rectal swab)
Compare rate of diarrhea | 7 days
  To compare the rate of diarrhea (≥ 4 loose stools within 24 hours) following administration of each vaccine regimen versus placebo over 7 days of follow-up

OTHER OUTCOMES:
Plot seroconversion | Day 7, 14, 21, 28, 35 and 42
  To plot the seroconversion (≥ 4-fold increase over baseline), mean fold rise (comparing baseline titer with post-vaccination titer), and kinetics of serum IgG cholera antitoxin antibody following the ingestion of a single oral dose of PXVX0200 (CVD 103-HgR) containing ≥2 x10E8 cfu or ≥2 x10E9 cfu versus Shanchol™.
Assess reactogenicity | For seven days after each dose of PXVX0200
  Assess tiredness, vomiting, loss of appetite, abdominal pain and headache

CONTACTS AND LOCATIONS:
Overall Officials: Milagritos D Tapia, MD, Principal Investigator — University of Maryland, College Park; Samba O Sow, MD, MS, Principal Investigator — Centre pour le Developpement des Vaccins - Mali
Locations (1):
- Centre pour le Développement des Vaccins, Mali (CVD-Mali), Bamako, Mali

REFERENCES:
- [Derived] Sow SO, Tapia MD, Chen WH, Haidara FC, Kotloff KL, Pasetti MF, Blackwelder WC, Traore A, Tamboura B, Doumbia M, Diallo F, Coulibaly F, Onwuchekwa U, Kodio M, Tennant SM, Reymann M, Lam DF, Gurwith M, Lock M, Yonker T, Smith J, Simon JK, Levine MM. Randomized, Placebo-Controlled, Double-Blind Phase 2 Trial Comparing the Reactogenicity and Immunogenicity of a Single Standard Dose to Those of a High Dose of CVD 103-HgR Live Attenuated Oral Cholera Vaccine, with Shanchol Inactivated Oral Vaccine as an Open-Label Immunologic Comparator. Clin Vaccine Immunol. 2017 Dec 5;24(12):e00265-17. doi: 10.1128/CVI.00265-17. Print 2017 Dec. PMID 29021299